CLINICAL TRIAL: NCT04117633
Title: Laparoscopic Suture Versus Mesh Rectopexy for the Treatment of Persistent Complete Rectal Prolapse in Children : A Comparative Randomized Study
Brief Title: Laparoscopic Suture Versus Mesh Rectopexy for the Treatment of Persistent Complete Rectal Prolapse in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, abdelaziz yehya, professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Azh-Ped-Surg-70712018
Record Dates: First submitted 2019-09-28; First posted 2019-10-07 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Rectal Prolapse
Keywords: Rectal Prolapse; Laparoscopy; Mesh; Rectopexy; pediatrics
MeSH Terms: conditions — Rectal Prolapse | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: The study included two equal groups. one group underwent laparoscopic mesh rectopexy and the other underwent suture rectopexy.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesh Rectopexy (Active Comparator): Using Laparoscopy
  Interventions: Device: Laparoscopy
- Suture Rectopexy (Active Comparator): Using Laparoscopy
  Interventions: Device: Laparoscopy

INTERVENTIONS:
Device: Laparoscopy — Laparoscopic Procedures for Rectopexy

SUMMARY:
Purpose: to compare Laparoscopic mesh rectopexy with laparoscopic suture rectopexy The operative time, recurrence rate, post-operative constipation, and effect on fecal incontinence, were reported and evaluated for each group Results:

DETAILED DESCRIPTION:
Purpose: to compare Laparoscopic mesh rectopexy with laparoscopic suture rectopexy Patient and Methods: The prospective study was conducted at Pediatric Surgery Department, Al-Azhar university hospitals, Cairo, Egypt . The operative time, recurrence rate, post-operative constipation, and effect on fecal incontinence, were reported and evaluated for each group

ELIGIBILITY:
Inclusion Criteria:

Children with persistant complete Rectal Prolapse.

* Failure of conservative treatment.
* more than 2 attacks of prolapse requiring manual reduction.

Exclusion Criteria:

* Sever constipation
* Previous abdominal or pelvic surgery with extensive adhesions.
* Cases older than 12ys,
* Patients with rectal polyp

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Signs of improvement | 12 weeks
  No recurrence of Rectal Prolapse

SECONDARY OUTCOMES:
Signs of improvement | 30 weeks
  Improvement of Fecal Incontinence score(Rintala score)